CLINICAL TRIAL: NCT07051161
Title: Impact of Interventional Endoscopy on Quality of Life in Patients With Acute Respiratory Distress Due to Tumor Compression or Obstruction of the Lower Respiratory Tract
Acronym: ENDoRA
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC24.0408; 2024-A02698-39 (Other: ID RCB)
Record Dates: First submitted 2025-06-12; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Solid Cancer; Bronchial Endoscopy; Therapeutic Bronchofiberscopy
MeSH Terms: interventions — Bronchoscopes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: bronchoscope — procedure performed by bronchoscopy
  Other Names: desobstruction of lower respiratory tract

SUMMARY:
Bronchoscopic endoscopy has shown its effectiveness and reliability for the treatment (desobstruction or prothesis) of tumor-induced bronchial obstructions, particularly in the first few weeks. The presence of a lower airway prosthesis can lead to device obstruction requiring daily inhaled fluidification, bacterial colonization, migration of the prosthesis, or the appearance of obstructive or hemorrhagic granulomas.

The aim of this study is to evaluate the quality of life of patients after endobronchial treatment.

It is a prospective, descriptive, and multicentric (national) study. The main objective is to compare the total score on the Saint-George questionnaire at J7 of the interventional endoscopy compared to before the procedure.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* tumoral tracheobronchial obstruction and/or compression
* proven solid cancer or suspicion
* Acute respiratory distress (at least one of the 5):

  * RR : ≥25/min
  * Sign of respiratory struggle
  * Sign of respiratory failure
  * Oxygen therapy ≥5L/min
  * Ventilatory support (NIV, OHD or IT) :
* Indication for therapeutic interventional endoscopy
* No guardianship or curatorship
* Non-hematological tumor

Exclusion Criteria:

* Minors
* patients with neurological disabilities unable to understand and respond to the questionnaire
* patients under guardianship or curatorship

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inclusion Criteria:
  * >18 years old
  * tumoral tracheobronchial obstruction and/or compression
  * proven solid cancer or suspicion
  * Acute respiratory distress (at least one of the 5):
    * RR : ≥25/min
    * Sign of respiratory struggle
    * Sign of respiratory failure
    * Oxygen therapy ≥5L/min
    * Ventilatory support (NIV, OHD or IT) :
  * Indication for therapeutic interventional endoscopy
  * No guardianship or curatorship
  * Non-hematological tumor
  Exclusion Criteria:
  * Minors
  * patients with neurological disabilities unable to understand and respond to the questionnaire
  * patients under guardianship or curatorship
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Saint George Score (quality of life) | At inclusion, and 7 days after therapeutic bronchoscopy
  Difference between Saint-George score at inclusion and Day 7.
  The scores for each dimension range from 0 to 100, with a score of 100 indicating excellent health.

SECONDARY OUTCOMES:
Saint-George and SF-12 (12-Item Short-Form Health Survey) score | at inclusion and Day 30
  Difference of these scores between inclusion and Day 30
  The scores for each dimension of the Saint-George score range from 0 to 100, with a score of 100 indicating excellent health.
  The SF-12 score ranges from 1 to 60, with a score of 60 indicating very poor quality of life.
ECOG-performance Status | inclusion and Day 30
  It ranges from 0 (fully active) to 5 (dead).
Duration of ventilatory support (mechanical ventilation, non-invasive ventilation, high-flow oxygen) | During the 30 first days from intervention
hospitalization duration | During the 30 first days from intervention
anti-tumoral treatment | During the 30 first days from intervention
  initiation or continuation of anti-tumour treatment (radiotherapy, chemotherapy, immunotherapy, targeted therapy)
survival | through study completion, an average of 1 year

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roy P, Fournier C, Barnestein R, Wallyn F, Bourinet V, Briault A, Camuset J, Cellerin L, Crutu A, Dewolf M, Egenod T, Favrolt N, Heluain V, Lorut C, Mangiapan G, Schlossmasscher P, Toublanc B, Usturoi D, Legodec J, Vergnon JM, Pajiep Chapda MC, Dutau H, Guibert N. Outcomes of Therapeutic Bronchoscopy in Malignant Airway Obstruction Causing Acute Respiratory Failure. Ann Am Thorac Soc. 2024 May;21(5):833-837. doi: 10.1513/AnnalsATS.202311-943RL. No abstract available. PMID 38391185
- [Background] Roy P, Roy P, Amari L, Laroumagne S, Legodec J, Fournier C, Cellerin L, Lorut C, Gonin F, Vergnon JM, Egenod T, Favrolt N, Schlossmacher P, Bourinet V, Perrot L, Lachkar S, Camuset J, Briault A, Degot T, Gut-Gobert C, Mangiapan G, Jasnot JY, Briens E, Crutu A, Marceau A, Toublanc B, Dewolf M, Dutilh J, Germain N, Tronchetti J, Astoul P, Guibert N, Dutau H. Predictive Factors of Clinical Success of Therapeutic Bronchoscopy in Malignant Central Airway Obstruction: Results from the EpiGETIF Registry. Respiration. 2025;104(9):667-677. doi: 10.1159/000545568. Epub 2025 Apr 4. PMID 40188807